CLINICAL TRIAL: NCT06597955
Title: Large-Scale Implementation of a Decision Aid About Colorectal Cancer Screening
Acronym: IDecide
Status: Enrolling by invitation | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other); Eskenazi Health (Other)
Responsible Party: Principal Investigator, Peter Schwartz, Principal Investigator, Indiana University
Other Study IDs: 22517; SDM-2022C2-28397 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer Screening
Keywords: decision aid; implementation; colorectal cancer; shared decision making; electronic health record
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare system leadership, providers, and staff: Leadership, providers, and staff at the project team's affiliated healthcare system
- Patients due for colorectal cancer screening: Patients who are considered due for colorectal cancer screening prior to a scheduled appointment with a primary care provider at the project team's affiliated healthcare system and completed the appointment.

SUMMARY:
The goal of the project is to improve shared decision making and increase uptake of colorectal cancer (CRC) screening by facilitating the implementation of a decision aid about CRC and screening options in two healthcare systems in Indiana.

DETAILED DESCRIPTION:
This implementation project is putting a shared decision making approach into routine practice to help patients make informed decisions about colorectal cancer(CRC) screening. Regular screening is recommended for adults ages 45 - 75 years old, and there are multiple approved tests for individuals at average risk for colorectal cancer. A video-based decision aid about CRC screening was developed and tested in a previous study by the project team. The study showed that viewing the decision aid had positive effects on measures directly related to shared decision making (knowledge, decision conflict) as well as intent to undergo CRC screening. The project team is working with two healthcare systems to provide patients who are eligible for CRC screening access to the decision aid, training staff and clinicians how to use the decision aid to support shared decision making for CRC screening, working with healthcare system leaders to support the staff and clinicians, and providing support for the ongoing use of the decision aid.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare system participants will be eligible if they are employed by one of the project team's partner healthcare systems
* Patient participants will be eligible if they are considered due for colorectal cancer screening by the healthcare systems' criteria.

Exclusion Criteria:

Patient participants will be excluded if they:

* are not between ages of 45 - 75 years old
* self-report that they no longer receive primary care at either of the project team's partner healthcare systems
* self-report that they are not due for colorectal cancer screening (had colonoscopy within the past 10 years, sigmoidoscopy in the last 5 years, FIT in the past year, or Cologuard in the past 3 years)
* are unable to speak or read English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will be healthcare system primary care patients, and health system leadership, clinicians, and staff involved in primary care.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Shared decision making | 18 months
  Shared decision making will be assessed using the CollaboRATE scale. CollaboRATE is a three-item measure that assesses three key areas of shared decision making; 1) explaining the health issue; 2) asking for patient preferences; and 3) incorporating patient preferences into the decision. Each item uses 0 - 9 likert response options ranging from 0 = "no effort was made" to 9 = "every effort was made". The higher the score the better the shared decision making.
Implementation of decision aid | 18 months
  Interviews with healthcare system leadership, clinicians, staff and patients

CONTACTS AND LOCATIONS:
Overall Officials: Peter H. Schwartz, MD, PhD, Principal Investigator — Indiana University; Teresa M. Damush, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States